CLINICAL TRIAL: NCT05670093
Title: Neural Pressure Support, a Randomized Crossover Trial
Brief Title: Neural Pressure Support, Synchrony and Respiratory Muscle Unloading
Acronym: NPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Francesca Campoccia Jalde, Francesca Campoccia Jalde, MD, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k 2021-5369
Record Dates: First submitted 2022-11-19; First posted 2023-01-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Intervention Model Description: Interventional prospective study. Each participant is ventilated both on PS and NPS at 3 different support levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neural Pressure Support (Experimental): Patients will be ventilated in Pressure Support and Neural Pressure Support at 3 different levels of support in randomized order
  Interventions: Device: Neural Pressure Support (mode of mechanical ventilation)

INTERVENTIONS:
Device: Neural Pressure Support (mode of mechanical ventilation) — Nasogastric tube will be removed and replaced by a Esophageal catheter and Electrical Diaphragm activity catheter and mechanical ventilation in mode Neural Pressure Support

SUMMARY:
In this study patients who are intubated and on ventilator for more than 24h will be ventilated at three different level of support in Pressure Support and Neural Pressure Support to study patient-ventilator synchrony and muscle unloading.

DETAILED DESCRIPTION:
This study is an interventional randomized crossover study in intubated and mechanically ventilated patients for more than 24h. Eligible patients from whom informed consent is obtained and Pes and Edi catheter are successfully positioned are enrolled in the study. Patients will be ventilated in Pressure Support and Neural Pressure Support at three different level of assist (baseline, 50% and 150% of baseline respectively) in randomized order. Ventilator curves will be recorded and bloodgas obtained at the end of each study step, each lasting 20min.

ELIGIBILITY:
Inclusion Criteria:

-Patients intubated for more than 24 hours in the weaning phase from the ventilator.

Exclusion Criteria:

* bleeding disorders (PK INR>1,5 or APTT>50s or platelet count <50000/µL)
* unstable circulation (requiring high vasopressor dose, for example Noradrenalin >0,2µg/kg/min)
* severe lung disease (PFI ≤ 13,3 kPa)
* fever> 38,5°C
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient-ventilator asynchronies | 20 minutes ventilatory traces recording
  quantification of asynchronies by the use of the Edi catheter

SECONDARY OUTCOMES:
respiratory muscle unloading | 20 minutes ventilatory traces recording
  quantification of muscle unloading by use of Pes

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Campoccia Jalde, Principal Investigator — Department of Molecular Medicine and Surgery, Karolinska Institutet, Stockholm, Sweden.
Locations (1):
- Karolinska University Hospital, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No